CLINICAL TRIAL: NCT01135446
Title: Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of Ultra Low Doses of Dapagliflozin in Healthy Subjects
Acronym: ULDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MB102-088
Record Dates: First submitted 2010-05-27; First posted 2010-06-02 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- dapagliflozin (0.001 mg) (Experimental): Cohort 1
  Interventions: Drug: dapagliflozin
- dapagliflozin (0.01 mg) (Experimental): Cohort 2
  Interventions: Drug: dapagliflozin
- dapagliflozin (0.1 mg) (Experimental): Cohort 3
  Interventions: Drug: dapagliflozin
- dapagliflozin (0.3 mg) (Experimental): Cohort 4
  Interventions: Drug: dapagliflozin
- dapagliflozin (1 mg) (Experimental): Cohort 5
  Interventions: Drug: dapagliflozin
- dapagliflozin (2.5 mg) (Experimental): Cohort 6
  Interventions: Drug: dapagliflozin

INTERVENTIONS:
Drug: dapagliflozin — Oral Solution, Oral, 0.001 mg, once on Day 1 only, 2 days
  Other Names: BMS-512148
  Arms: dapagliflozin (0.001 mg)
Drug: dapagliflozin — Oral Solution, Oral, 0.01 mg, once on Day 1 only, 2 days
  Other Names: BMS-512148
  Arms: dapagliflozin (0.01 mg)
Drug: dapagliflozin — Oral Solution, Oral, 0.1 mg, once on Day 1 only, 2 days
  Other Names: BMS-512148
  Arms: dapagliflozin (0.1 mg)
Drug: dapagliflozin — Tablets, Oral, 0.3 mg, once on Day 1 only, 2 days
  Other Names: BMS-512148
  Arms: dapagliflozin (0.3 mg)
Drug: dapagliflozin — Tablets, Oral, 1 mg, once on Day 1 only, 2 days
  Other Names: BMS-512148
  Arms: dapagliflozin (1 mg)
Drug: dapagliflozin — Tablets, Oral, 2.5 mg, once on Day 1 only, 2 days
  Other Names: BMS-512148
  Arms: dapagliflozin (2.5 mg)

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamics (PD), pharmacokinetics (PK), safety and tolerability following single oral doses of 0.001 mg to 2.5 mg dapagliflozin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* WOCBP who are using acceptable method of contraception
* Women who are not nursing

Exclusion Criteria:

* History of GI disease
* Any GI surgery that could impact study drug absorption
* Glucosuria at screening or Day -2
* Abnormal liver function tests (ALT, AST or total bilirubin > 10% above ULN)
* History of current or recurrent UTI
* History of Diabetes Mellitus
* History of chronic or recurrent vulvovaginal mycotic infections
* Estimated creatinine clearance (ClCr) < 80 mL/min using Cockroft-Gault formula
* History of allergy to SGLT2 inhibitors or related compounds

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Total 24-hour Urinary Glucose Excretion as a Measure of Pharmacodynamic Effect | 24 hours after dosing

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 hours after dosing
Dapagliflozin and Dapagliflozin 3-O-glucuronide (Metabolite of Dapagliflozin) Concentrations to Characterize Dapagliflozin Pharmacokinetics | 2 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Lp, Austin, Texas, United States

REFERENCES:
- See also: MB102-088_redacted_CSR_synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3653&filename=MB102-088_redacted_CSR_synopsis.pdf